CLINICAL TRIAL: NCT02652026
Title: Effect of Non-surgical Periodontal Treatment on HbA1c in Type 2 Diabetic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Responsible Party: Principal Investigator, elisabet mauri i obradors, Dentistry, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UBarcelona
Record Dates: First submitted 2015-07-11; First posted 2016-01-11 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Chronic Periodontitis; Type 2 Diabetes Mellitus
Keywords: dental root planing and scaling; periodontal disease; type 2 diabetes mellitus; glycosylated hemoglobin A
MeSH Terms: conditions — Chronic Periodontitis; Diabetes Mellitus, Type 2; Periodontal Diseases | interventions — Tooth Exfoliation; Root Planing; Dental Prophylaxis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment Group (Experimental): The Treatment Group (TG) received full mouth debridement, which consisted of scaling and root planing (SRP), was done in a single visit using an ultrasonic scaler (SATELEC P5 Newtron, Acteon, Merignac, France) and Gracey curettes (Hu- Friedy, Chicago, USA).Also received Oral Hygienic Instructions
  Interventions: Procedure: Nonsurgical periodontal treatment; Procedure: Dental Prophylaxis
- Control Group (Active Comparator): The Control Group (CG) received periodontal prophylaxis at baseline, by removal of supragingival deposits (plaque and calculus) with ultrasonic scaler. Also received Oral Hygienic Instructions
  Interventions: Procedure: Dental Prophylaxis

INTERVENTIONS:
Procedure: Nonsurgical periodontal treatment — Full mouth debridement, which consisted of scaling and root planing (SRP), was done in a single visit using an ultrasonic scaler (SATELEC P5 Newtron XS, Acteon, Merignac, France) and Gracey curretes (Hu- Friedy, Chicago, USA).
  Other Names: Scaling and root planing
  Arms: Treatment Group
Procedure: Dental Prophylaxis — Removal superficial plaque using an ultrasonic scaler (SATELEC P5 Newtron XS, Acteon, Merignac, France)
  Other Names: Removal superficial plaque

SUMMARY:
The main objective is to evaluate the effect of nonsurgical periodontal treatment on serum levels of HbA1c in patients with type 2 diabetes mellitus (T2DM). This study is a 6-month, single-masked, randomized clinical trial.A total of 90 patients with diabetes and chronic generalized periodontal disease will be randomly divided into 2 groups: Treatment Group, Control Group.

DETAILED DESCRIPTION:
Background: Periodontitis and diabetes are both highly prevalent conditions, and the association between these two common diseases has been recognised by dental professionals for many years.

Aim: The main objective is to evaluate the effect of nonsurgical periodontal treatment on serum levels of HbA1c in patients with type 2 diabetes mellitus (T2DM).

Methods: This study is a 6-month, single-masked, randomized clinical trial.A total of 90 patients with diabetes and chronic generalized periodontal disease will be randomly divided into 2 groups: Treatment Group (TG) (Oral Hygiene Instructions (OHI) + scaling and root planing (RAR) using ultrasound device and Gracey curettes); Control Group (CG) (OHI + supragingival removal of plaque and calculus with ultrasonic device). CG patients receive salvage therapy if a significant worsening of their periodontal status and / or metabolic observed. Periodontal assesment (probing pocket depth (PPD), gingival index (GI), and plaque index (PI)) and systemic assesment (random blood sugar, glycosylated hemoglobin (HbA1C), and salivary cytokines) and bacterial asessment at baseline and 3, 6 months after treatment is performed. There will be a single examiner, blind and calibrated to improve reproducibility. The investigators' hypothesis is that non-surgical periodontal treatment reduces HbA1c, improving metabolic control in patients with DM

ELIGIBILITY:
Inclusion criteria were:

* Diagnostic of T2DM (diagnosed at least 1'5 years prior the study).
* Presence of generalized chronic periodontitis (With at least 9 teeth present and more than 30% of locations with probing depth (PD) and clinical attachment level (CAL) ≥4mm).

Exclusion criteria included:

* Patients who received antibiotics the last 15 days, or for a period longer than 10 days the last three months.
* Having received non-surgical periodontal treatment within the past 6 months.
* Pregnancy
* Significant change of medication for diabetes during the course of the study
* Evidence of other serious systemic disease (ASA III or IV) which may influence periodontal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Glycosylated Hemoglobin (HbA1c) | Baseline and 6 months after intervention
  Serum levels glycosylated hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Jose López-López, Phd, Study Director — University of Barcelona